CLINICAL TRIAL: NCT02644746
Title: Efficacy and Safety of Acupuncture for Degenerative Lumbar Spinal Stenosis: Protocol for a Randomized Placebo-controlled Trial
Brief Title: Efficacy and Safety of Acupuncture for Degenerative Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Qin Zongshi, Dr., Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015EC114
Record Dates: First submitted 2015-12-27; First posted 2016-01-01 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Degenerative Lumbar Spinal Stenosis
Keywords: degenerative lumbar spinal stenosis; acupuncture; randomized controlled trial
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture group (Experimental): Acupuncture has a long time used for chronic pain including low back pain, sciatica, and other pain related to spina via stimulating specific acupuncture points.
  Interventions: Device: acupuncture
- Placebo needle group (Placebo Comparator): The placebo needle using in this trial will be unpenetrated needles. Based on our previous research, the placebo needle is a valid control for acupuncture research and may eliminate the placebo effect of acupuncture.
  Interventions: Device: placebo needle

INTERVENTIONS:
Device: acupuncture — Shenshu (BL23), Dachangshu (BL25), Weizhong (BL40), Chengshan (BL57), Taixi (KI3) acupoints will be used. For bilateral Dachangshu (BL 25), the needle will be inserted vertically at approximately 40-70 mm until participants got a electric shock feeling downward to calves, then the needle should be elevated up 2 mm, without rotating or lifting. For other four acupoints (BL23, BL40, BL57, KI3), they will be inserted 10 to 15 mm in depth with three times light amplitude rotation and lift to induce a sensation of soreness. The manipulations will be performed 3 times in total during 1 session (every 10 min). There are 24 treatment sessions after baseline, 3 times a week, and the patients will undergo a 30-min treatment each session.
  Arms: Acupuncture group
Device: placebo needle — Acupuncturists will use blunt tip needles (Huatuo, Suzhou, China) that cannot penetrate skin and stimulate deep tissues, and the thrusting and twisting motions will be used by acupuncturists to simulate the treatment and blind the patients. Each placebo needle consists of four parts: needle handle, needle body, blunt tip and adhesive pad. The chosen of acupoints, treatment duration, and frequency of sessions will be the same as the acupuncture group. To guarantee blinding, the investigators will make appointments with each participant on alternate days to prevent crosstalk among groups.
  Arms: Placebo needle group

SUMMARY:
Degenerative Lumbar spinal stenosis (DLSS) is a major problem for public health and the primary reason the older seek lumbar spine surgery. Acupuncture is safe and maybe effective for DLSS but the evidence is poor. Therefore, an objective assessment of acupuncture efficacy is critical for making informed decisions about its appropriate role for patients. A total of 80 participants meet prior inclusion criteria will be recruited. The participants will be allocated to acupuncture group or placebo needle (unpenetrated acupuncture) group randomly. Twenty-four treatments will be provided over 8 weeks. The primary change of Modified Roland-Morris Disability Questionnaire (RMDQ) and secondary outcomes including the change of Number Rating Scale (NRS); the change of Self-paced Walking test (SPWT); the change of Swiss Spinal Stenosis Questionnaire (SSSQ); the expectations that acupuncture might help participants with DLSS. All outcomes will be assessed at baseline, and/or after 4, 8, 20 and 32 weeks. Statistical analysis will include independent sample t-test, Chi-squared test and non-parametric test. The investigators hope the result of this trial will clarify the value of acupuncture for DLSS and help clinicians make proper decisions.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following conditions will be considered for enrollment. The inclusion criteria are as follows:

1. Pain in the low back, buttock, and/or lower extremity with standing, walking and/or spinal extension. (Using NRS questionnaire to measure pain symptoms, and pain measured by NRS ≥ 4.)
2. Roland-Morris score of at least 7.
3. Mild-moderate-severe lumbar central canal spinal stenosis identified by MRI or CT scan.
4. Lower extremity symptoms consistent with neurogenic claudication.
5. Age 50 to 80 years old.
6. Signed the consent and take part in this trial of his/her willing.

Exclusion Criteria:

1. Congenital stenosis of vertebral canal, serious indications of DLSS (such as segmental muscular atrophy, bowel and bladder disturbances), spinal nerve root canal stenosis, lumbar spondylolysis, lumbar tuberculosis, lumbar vertebral tumors, and vertebral body compression fracture.
2. Spinal instability requiring surgery.
3. Severe vascular, pulmonary or coronary artery disease that limits ambulation including recent myocardial infarction.
4. Participants who have cognitive impairment that may render the subject unable to give informed consent or provide accurate data.
5. Clinical co-morbidities that could interfere with the collection of data concerning pain and function.
6. Acupuncture within the past 30 days.
7. Administered pain control drugs during the week prior to the baseline assessment (e.g.,non-steroidal anti-inflammatory drugs or herbal anti-inflammatory agents).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The change of Modified Roland-Morris Disability Questionnaire (RMDQ) from baseline. | Baseline, week 1-4, week 5-8, week 9-20, week 21-32

SECONDARY OUTCOMES:
The change of Number Rating Scale (NRS) from baseline. | Baseline, week1-8, week 9-20, week 21-32
The change of Self-paced Walking test (SPWT) from baseline to week 8. | Baseline, week 8.
The change of Swiss Spinal Stenosis Questionnaire (SSSQ) from baseline. | Baseline, week 1-4, week 5-8, week 9-20, week 21-32
The expectations that acupuncture might help patients DLSS will be recorded at baseline (scale). | Baseline.
  This expectation scale include four items, including belief "Do you think acupuncture can work?", expectation "Do you think acupuncture may help your "DLSS", preference 1"Which treatment do you prefer?", and preference2 "Did you get your treatment preference?" In fact, this is partial domain of "participants baseline information", which will be recorded at baseline. The investigators want to explore the relationship between expectation degree and primary outcome via linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be preserved, when the paper submitted, if the journal ask IPD, it will be uploaded as a supplement.

REFERENCES:
- [Derived] Qin Z, Ding Y, Wu J, Zhou J, Yang L, Liu X, Liu Z. Efficacy of acupuncture for degenerative lumbar spinal stenosis: protocol for a randomised sham acupuncture-controlled trial. BMJ Open. 2016 Nov 16;6(11):e012821. doi: 10.1136/bmjopen-2016-012821. PMID 27852717